CLINICAL TRIAL: NCT05164120
Title: A Proof of Concept, Randomized, Double-blind, Placebo-controlled Trial of Orally Administered Belnacasan Tablets for the Treatment of Mild to Moderate COVID-19
Brief Title: Safety, Tolerability, and Treatment Effect of Belnacasan in Patients With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedStar Health (Other)
Responsible Party: Sponsor
Organization: Medstar Health Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MedStar-COVID-19-belnacasan
Record Dates: First submitted 2021-12-15; First posted 2021-12-20 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — belnacasan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomizations, assigned 1:1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): 900mg dose TID Administration Total: 2700mg
  Interventions: Drug: Belnacasan
- Placebo (Placebo Comparator): 0 mg dose TID Administration Total: 0 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Belnacasan — Oral administration
  Arms: Interventional
Drug: Placebo — Tablet containing 0mg of API
  Arms: Placebo

SUMMARY:
The purpose of this trial is to assess the safety, tolerability and treatment effect of the orally administered Caspase-1 inhibitor, belnacasan, for the treatment of patients with mild to moderate COVID-19 and to generate proof of concept for future trials.

DETAILED DESCRIPTION:
COVID-19 is an acute respiratory disease caused by the SARS-CoV-2 virus which has impacted the lives of millions of patients. Though vaccines and preventive treatments such as monoclonal antibodies, steroids, and anti-virals have been established, they do not specifically target the resulting inflammatory response and complications the virus causes.

This study aims to evaluate how safe and effective a particular oral medication, Belnacasan, is in diminishing your body's inflammatory response, which may go into overdrive when infected with the virus. This overly activated immune response can become uncontrolled resulting in cell death and the release of damaging proteins which can cause major harm to all organs throughout the body.

Belnacasan prevents the activation of a particular enzyme, Caspase-1, which plays a major role in activating this damaging immune response brought on by COVID-19. The goal of this medication being a more targeted treatment that aims to prevent the devastating immune response.

ELIGIBILITY:
Inclusion Criteria:

1. Subject (or legally authorized representative) provides written informed consent prior to the initiation of any study procedures
2. Subject understands and agrees to comply with planned study procedures, including using the diary
3. Subject agrees to the collection of nasopharyngeal swabs and venous blood per protocol
4. Subject is male or non-pregnant female adult ≥18 years of age at time of consent

   a. Women with a history of menstruation must agree to use two methods of contraception, at least one of which is highly effective, for the duration of the study as well as to undergo additional pregnancy testing during the study
5. Subject has a laboratory confirmed SARS-CoV-2 infection as determined by RT-PCR assay prior to enrollment
6. Subject has evidence of either mild or moderate COVID-19 illness of less than 7 days from first onset, with minimal baseline symptom severity based on patient-reported FDA scoring system defined as follows:

   1. Subject presents with at least two common symptoms of COVID-19 from the following list: Stuffy or runny nose, sore throat, cough, low energy or tiredness, muscle or body ache, headache, chills or shivering, feeling hot or feverish, nausea, vomiting, diarrhea, shortness of breath with exertion (without supplemental oxygen requirement) with a score of 2 or higher, impairment in sense of smell or taste with a score of 1 or higher OR
   2. Subject presents with any (i.e., at least one) symptom of COVID-19 as defined above AND clinical evidence of moderate COVID-19 as defined by FDA guidance for industry (such as respiratory rate >20 breaths per minute, heart rate >90 beats per minute, with oxygen saturation >93% on room air at sea level)
7. Subject presents with high-risk for COVID-19-related inflammation determined by at least one comorbidity, including obesity, diabetes, hypertension, stable heart disease, respiratory disease, and/or non-severe fatty liver disease
8. Subject's overall health condition is deemed as suitable to fully and safely participate in this trial as determined by the investigator

Exclusion Criteria:

1. Any clinical signs indicative of severe or critical COVID-19 as defined by FDA guidance for Industry at the time, including SpO2 <93% and/or oxygen requirement
2. Hospitalization for COVID-19, or consideration thereof
3. ICU level of care and/or non-mechanical/mechanical ventilation and/or oxygen supplementation at time of enrollment
4. Pregnant or breast-feeding subjects
5. Subjects who cannot swallow tablets
6. History of any pre-existing organ impairment, such as:

   1. Severe kidney disease (known or estimated GFR <30 mL/minute) or on dialysis
   2. Uncontrolled, clinically significant heart diseases such as arrhythmias, angina or heart failure as defined by AHA/ACC Grade C and D
   3. Chronic respiratory disease requiring supplemental oxygen
   4. Moderate and severe hepatic impairment as defined by Child-Pugh scoring Class B and Class C
7. Elevated liver function test (determined by ALT, AST, GGT, or ALP >2x upper limit of normal, and/or total Bilirubin > upper limit of normal)
8. History of malignancy or immunodeficiency within the prior 5 years
9. Acute respiratory illness other than COVID-19
10. Acute bacterial, viral or fungal infection (including HIV, hepatitis B, hepatitis C)
11. While dosed with IP, the taking of prohibited concomitant medication or the ingestion of food that interferes with the IP, including:

    1. Non-COVID19-related anti-viral medication such as lopinavir, ritonavir, ribavirin, or interferon-1β
    2. Systemically administered immunosuppressive and anti-inflammatory agents, other than background standard of care for COVID-19 at the time
    3. Drugs and foods that are potent inhibitors or inducers of CYP3A4 and/or P-gp, as listed in FDA "Drug Development and Drug Interactions: Table of Substrates, Inhibitors and Inducers", including herbal medications such as St. John's Wort within 30 days or 5 half-lives (whichever is longer) prior to the first dose of study drug
12. Any other diseases or medical conditions or concomitant medications that are deemed as not compatible or appropriate for the subject's ability to fully and safely participate in this trial as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Wortmann, MD, Principal Investigator — MedStar Health
Locations (2):
- United States (2):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - MedStar Franklin Square, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 0 mg dose TID Administration Total: 0mg
  Placebo: Tablet containing 0mg of API
Period: Overall Study
Arm/Group | Interventional | Placebo
Started | 20 | 20
Completed | 18 | 18
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interventional | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (11.9) | 41.6 (12.1) | 43.4 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 13 | 11 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Belnacasan
Description: Number of adverse events and serious adverse events
Time Frame: Through 60 days post enrollment
Population: Patients reporting AEs and SAEs from the time of enrollment through Day 60
Measure: Number; unit: Number of AEs and SAEs
Arm/Group | Interventional | Placebo
Number analyzed (Participants) | 20 | 20
Number of AEs and SAEs
  Number of adverse events | 11 | 10
  Number of serious adverse events | 0 | 0

2. Secondary Outcome: Sustained Recovery and Resolution Rates of Common COVID-19 Symptoms
Description: Proportion of subjects in treatment group versus placebo group, respectively, who, per symptom questionnaire, rate stuffy or runny nose, sore throat, cough, low energy or tiredness, muscle or body ache, headache, chills or shivering, feeling hot or feverish, nausea, vomiting, diarrhea, shortness of breath at rest, shortness of breath with exertion, or impairment in sense of smell or taste as mild, moderate or severe.
Time Frame: Baseline and Days 4, 7, 10, 14, 21, 28, 42, and 60 post randomization
Population: Proportion of subjects in treatment group versus placebo group, respectively, who, per symptom questionnaire, rate stuffy or runny nose, sore throat, cough, low energy or tiredness, muscle or body ache, headache, chills or shivering, feeling hot or feverish, nausea, vomiting, diarrhea, shortness of breath at rest, shortness of breath with exertion, or impairment in sense of smell or taste ranging from mild to moderate.
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional | Placebo
Number analyzed (Participants) | 20 | 20
Participants
  Runny/stuffy nose at Baseline | 14 | 19
  Runny/stuffy nose at Day 4: number analyzed (Participants) | 19 | 19
  Runny/stuffy nose at Day 4 | 13 | 13
  Runny/stuffy nose at Day 7: number analyzed (Participants) | 18 | 19
  Runny/stuffy nose at Day 7 | 17 | 17
  Runny/stuffy nose at Day 10: number analyzed (Participants) | 18 | 19
  Runny/stuffy nose at Day 10 | 6 | 4
  Runny/stuffy nose at Day 14: number analyzed (Participants) | 18 | 18
  Runny/stuffy nose at Day 14 | 12 | 10
  Runny/stuffy nose at Day 21: number analyzed (Participants) | 16 | 18
  Runny/stuffy nose at Day 21 | 5 | 3
  Runny/stuffy nose at Day 28: number analyzed (Participants) | 18 | 18
  Runny/stuffy nose at Day 28 | 5 | 1
  Runny/stuffy nose at Day 42: number analyzed (Participants) | 17 | 18
  Runny/stuffy nose at Day 42 | 1 | 0
  Runny/stuffy nose at Day 60: number analyzed (Participants) | 17 | 17
  Runny/stuffy nose at Day 60 | 1 | 0
  Sore throat at Baseline | 13 | 14
  Sore throat at Day 4: number analyzed (Participants) | 19 | 19
  Sore throat at Day 4 | 4 | 3
  Sore throat at Day 7: number analyzed (Participants) | 18 | 19
  Sore throat at Day 7 | 14 | 9
  Sore throat at Day 10: number analyzed (Participants) | 18 | 19
  Sore throat at Day 10 | 1 | 0
  Sore throat at Day 14: number analyzed (Participants) | 18 | 18
  Sore throat at Day 14 | 4 | 2
  Sore throat at Day 21: number analyzed (Participants) | 16 | 18
  Sore throat at Day 21 | 0 | 0
  Sore throat at Day 28: number analyzed (Participants) | 18 | 18
  Sore throat at Day 28 | 1 | 0
  Sore throat at Day 42: number analyzed (Participants) | 17 | 18
  Sore throat at Day 42 | 0 | 0
  Sore throat at Day 60: number analyzed (Participants) | 17 | 17
  Sore throat at Day 60 | 0 | 0
  Cough at Baseline | 17 | 18
  Cough at Day 4: number analyzed (Participants) | 19 | 19
  Cough at Day 4 | 13 | 12
  Cough at Day 7: number analyzed (Participants) | 18 | 19
  Cough at Day 7 | 16 | 18
  Cough at Day 10: number analyzed (Participants) | 18 | 19
  Cough at Day 10 | 7 | 9
  Cough at Day 14: number analyzed (Participants) | 18 | 18
  Cough at Day 14 | 11 | 15
  Cough at Day 21: number analyzed (Participants) | 16 | 18
  Cough at Day 21 | 7 | 6
  Cough at Day 28: number analyzed (Participants) | 18 | 18
  Cough at Day 28 | 6 | 3
  Cough at Day 42: number analyzed (Participants) | 17 | 18
  Cough at Day 42 | 1 | 0
  Cough at Day 60: number analyzed (Participants) | 17 | 17
  Cough at Day 60 | 1 | 0
  Low energy or tiredness at Baseline | 17 | 14
  Low energy or tiredness at Day 4: number analyzed (Participants) | 19 | 19
  Low energy or tiredness at Day 4 | 10 | 7
  Low energy or tiredness at Day 7: number analyzed (Participants) | 18 | 19
  Low energy or tiredness at Day 7 | 18 | 17
  Low energy or tiredness at Day 10: number analyzed (Participants) | 18 | 19
  Low energy or tiredness at Day 10 | 6 | 1
  Low energy or tiredness at Day 14: number analyzed (Participants) | 18 | 18
  Low energy or tiredness at Day 14 | 11 | 4
  Low energy or tiredness at Day 21: number analyzed (Participants) | 16 | 18
  Low energy or tiredness at Day 21 | 6 | 3
  Low energy or tiredness at Day 28: number analyzed (Participants) | 18 | 18
  Low energy or tiredness at Day 28 | 7 | 1
  Low energy or tiredness at Day 42: number analyzed (Participants) | 17 | 18
  Low energy or tiredness at Day 42 | 1 | 0
  Low energy or tiredness at Day 60: number analyzed (Participants) | 17 | 17
  Low energy or tiredness at Day 60 | 0 | 0
  Muscle or body aches at Baseline | 13 | 11
  Muscle or body aches at Day 4: number analyzed (Participants) | 19 | 19
  Muscle or body aches at Day 4 | 7 | 1
  Muscle or body aches at Day 7: number analyzed (Participants) | 18 | 19
  Muscle or body aches at Day 7 | 13 | 13
  Muscle or body aches at Day 10: number analyzed (Participants) | 18 | 19
  Muscle or body aches at Day 10 | 2 | 0
  Muscle or body aches at Day 14: number analyzed (Participants) | 18 | 18
  Muscle or body aches at Day 14 | 6 | 1
  Muscle or body aches at Day 21: number analyzed (Participants) | 16 | 18
  Muscle or body aches at Day 21 | 3 | 2
  Muscle or body aches at Day 28: number analyzed (Participants) | 18 | 18
  Muscle or body aches at Day 28 | 3 | 0
  Muscle or body aches at Day 42: number analyzed (Participants) | 17 | 18
  Muscle or body aches at Day 42 | 1 | 0
  Muscle or body aches at Day 60: number analyzed (Participants) | 17 | 17
  Muscle or body aches at Day 60 | 0 | 0
  Headache at Baseline | 10 | 12
  Headache at Day 4: number analyzed (Participants) | 19 | 19
  Headache at Day 4 | 5 | 2
  Headache at Day 7: number analyzed (Participants) | 18 | 19
  Headache at Day 7 | 15 | 11
  Headache at Day 10: number analyzed (Participants) | 18 | 19
  Headache at Day 10 | 4 | 1
  Headache at Day 14: number analyzed (Participants) | 18 | 18
  Headache at Day 14 | 5 | 5
  Headache at Day 21: number analyzed (Participants) | 16 | 18
  Headache at Day 21 | 3 | 1
  Headache at Day 28: number analyzed (Participants) | 18 | 18
  Headache at Day 28 | 5 | 2
  Headache at Day 42: number analyzed (Participants) | 17 | 18
  Headache at Day 42 | 2 | 0
  Headache at Day 60: number analyzed (Participants) | 17 | 17
  Headache at Day 60 | 0 | 0
  Chills or shivering at Baseline | 7 | 4
  Chills or shivering at Day 4: number analyzed (Participants) | 19 | 19
  Chills or shivering at Day 4 | 1 | 1
  Chills or shivering at Day 7: number analyzed (Participants) | 18 | 19
  Chills or shivering at Day 7 | 6 | 7
  Chills or shivering at Day 10: number analyzed (Participants) | 18 | 19
  Chills or shivering at Day 10 | 0 | 0
  Chills or shivering at Day: number analyzed (Participants) | 18 | 18
  Chills or shivering at Day | 1 | 1
  Chills or shivering at Day 21: number analyzed (Participants) | 16 | 18
  Chills or shivering at Day 21 | 1 | 0
  Chills or shivering at Day 28: number analyzed (Participants) | 18 | 18
  Chills or shivering at Day 28 | 2 | 0
  Chills or shivering at Day 42: number analyzed (Participants) | 17 | 18
  Chills or shivering at Day 42 | 0 | 0
  Chills or shivering at Day 60: number analyzed (Participants) | 17 | 17
  Chills or shivering at Day 60 | 0 | 0
  Feeling hot or feverish at Baseline | 8 | 8
  Feeling hot or feverish at Day 4: number analyzed (Participants) | 19 | 19
  Feeling hot or feverish at Day 4 | 3 | 0
  Feeling hot or feverish at Day 7: number analyzed (Participants) | 18 | 19
  Feeling hot or feverish at Day 7 | 10 | 10
  Feeling hot or feverish at Day 10: number analyzed (Participants) | 18 | 19
  Feeling hot or feverish at Day 10 | 0 | 0
  Feeling hot or feverish at Day 14: number analyzed (Participants) | 18 | 18
  Feeling hot or feverish at Day 14 | 1 | 1
  Feeling hot or feverish at Day 21: number analyzed (Participants) | 16 | 18
  Feeling hot or feverish at Day 21 | 0 | 0
  Feeling hot or feverish at Day 28: number analyzed (Participants) | 18 | 18
  Feeling hot or feverish at Day 28 | 1 | 0
  Feeling hot or feverish at Day 42: number analyzed (Participants) | 17 | 18
  Feeling hot or feverish at Day 42 | 0 | 0
  Feeling hot or feverish at Day 60: number analyzed (Participants) | 17 | 17
  Feeling hot or feverish at Day 60 | 0 | 0
  Nausea at Baseline | 6 | 1
  Nausea at Day 4: number analyzed (Participants) | 19 | 19
  Nausea at Day 4 | 2 | 1
  Nausea at Day 7: number analyzed (Participants) | 18 | 19
  Nausea at Day 7 | 7 | 3
  Nausea at Day 10: number analyzed (Participants) | 18 | 19
  Nausea at Day 10 | 2 | 0
  Nausea at Day 14: number analyzed (Participants) | 18 | 18
  Nausea at Day 14 | 3 | 1
  Nausea at Day 21: number analyzed (Participants) | 16 | 18
  Nausea at Day 21 | 0 | 2
  Nausea at Day 28: number analyzed (Participants) | 18 | 18
  Nausea at Day 28 | 2 | 0
  Nausea at Day 42: number analyzed (Participants) | 17 | 18
  Nausea at Day 42 | 0 | 0
  Nausea at Day 60: number analyzed (Participants) | 17 | 17
  Nausea at Day 60 | 0 | 0
  Vomiting at Baseline | 0 | 0
  Vomiting at Day 4: number analyzed (Participants) | 19 | 19
  Vomiting at Day 4 | 0 | 0
  Vomiting at Day 7: number analyzed (Participants) | 18 | 19
  Vomiting at Day 7 | 0 | 0
  Vomiting at Day 10: number analyzed (Participants) | 18 | 19
  Vomiting at Day 10 | 0 | 0
  Vomiting at Day 14: number analyzed (Participants) | 18 | 18
  Vomiting at Day 14 | 0 | 0
  Vomiting at Day 21: number analyzed (Participants) | 16 | 18
  Vomiting at Day 21 | 0 | 0
  Vomiting at Day 28: number analyzed (Participants) | 18 | 18
  Vomiting at Day 28 | 0 | 0
  Vomiting at Day 42: number analyzed (Participants) | 17 | 18
  Vomiting at Day 42 | 0 | 0
  Vomiting at Day 60: number analyzed (Participants) | 17 | 17
  Vomiting at Day 60 | 0 | 0
  Diarrhea at Baseline | 3 | 1
  Diarrhea at Day 4: number analyzed (Participants) | 19 | 19
  Diarrhea at Day 4 | 6 | 4
  Diarrhea at Day 7: number analyzed (Participants) | 18 | 19
  Diarrhea at Day 7 | 10 | 6
  Diarrhea at Day 10: number analyzed (Participants) | 18 | 19
  Diarrhea at Day 10 | 3 | 0
  Diarrhea at Day 14: number analyzed (Participants) | 18 | 18
  Diarrhea at Day 14 | 7 | 3
  Diarrhea at Day 21: number analyzed (Participants) | 16 | 18
  Diarrhea at Day 21 | 4 | 3
  Diarrhea at Day 28: number analyzed (Participants) | 18 | 18
  Diarrhea at Day 28 | 5 | 2
  Diarrhea at Day 42: number analyzed (Participants) | 17 | 18
  Diarrhea at Day 42 | 0 | 0
  Diarrhea at Day 60: number analyzed (Participants) | 17 | 17
  Diarrhea at Day 60 | 0 | 0
  Shortness of breath at rest at Baseline | 6 | 1
  Shortness of breath at rest at Day 4: number analyzed (Participants) | 19 | 19
  Shortness of breath at rest at Day 4 | 4 | 2
  Shortness of breath at rest at Day 7: number analyzed (Participants) | 18 | 19
  Shortness of breath at rest at Day 7 | 0 | 0
  Shortness of breath at rest at Day 10: number analyzed (Participants) | 18 | 19
  Shortness of breath at rest at Day 10 | 2 | 0
  Shortness of breath at rest at Day 14: number analyzed (Participants) | 18 | 18
  Shortness of breath at rest at Day 14 | 4 | 1
  Shortness of breath at rest at Day 21: number analyzed (Participants) | 16 | 18
  Shortness of breath at rest at Day 21 | 2 | 0
  Shortness of breath at rest at Day 28: number analyzed (Participants) | 18 | 18
  Shortness of breath at rest at Day 28 | 2 | 0
  Shortness of breath at rest at Day 42: number analyzed (Participants) | 17 | 18
  Shortness of breath at rest at Day 42 | 0 | 0
  Shortness of breath at rest at Day 60: number analyzed (Participants) | 17 | 17
  Shortness of breath at rest at Day 60 | 0 | 0
  Shortness of breath with exertion at Baseline | 7 | 5
  Shortness of breath with exertion at Day 4: number analyzed (Participants) | 19 | 19
  Shortness of breath with exertion at Day 4 | 5 | 4
  Shortness of breath with exertion at Day 7: number analyzed (Participants) | 18 | 19
  Shortness of breath with exertion at Day 7 | 14 | 10
  Shortness of breath with exertion at Day 10: number analyzed (Participants) | 18 | 19
  Shortness of breath with exertion at Day 10 | 5 | 3
  Shortness of breath with exertion at Day 14: number analyzed (Participants) | 18 | 18
  Shortness of breath with exertion at Day 14 | 8 | 2
  Shortness of breath with exertion at Day 21: number analyzed (Participants) | 16 | 18
  Shortness of breath with exertion at Day 21 | 4 | 2
  Shortness of breath with exertion at Day 28: number analyzed (Participants) | 18 | 18
  Shortness of breath with exertion at Day 28 | 2 | 1
  1Shortness of breath with exertion at Day 42: number analyzed (Participants) | 17 | 18
  1Shortness of breath with exertion at Day 42 | 1 | 1
  Shortness of breath with exertion at Day 60: number analyzed (Participants) | 17 | 17
  Shortness of breath with exertion at Day 60 | 0 | 1
  Impairment of sense of smell at Baseline | 4 | 3
  Impairment of sense of smell at Day 4: number analyzed (Participants) | 19 | 19
  Impairment of sense of smell at Day 4 | 4 | 3
  Impairment of sense of smell at Day 7: number analyzed (Participants) | 18 | 19
  Impairment of sense of smell at Day 7 | 5 | 5
  Impairment of sense of smell at Day 10: number analyzed (Participants) | 18 | 19
  Impairment of sense of smell at Day 10 | 1 | 1
  Impairment of sense of smell at Day 14: number analyzed (Participants) | 18 | 18
  Impairment of sense of smell at Day 14 | 1 | 2
  Impairment of sense of smell at Day 21: number analyzed (Participants) | 16 | 18
  Impairment of sense of smell at Day 21 | 1 | 1
  Impairment of sense of smell at Day 28: number analyzed (Participants) | 18 | 18
  Impairment of sense of smell at Day 28 | 0 | 0
  Impairment of sense of smell at Day 42: number analyzed (Participants) | 17 | 18
  Impairment of sense of smell at Day 42 | 0 | 0
  Impairment of sense of smell at Day 60: number analyzed (Participants) | 17 | 17
  Impairment of sense of smell at Day 60 | 0 | 0
  Impairment of sense of taste at Baseline | 6 | 6
  Impairment of sense of taste at Day 4: number analyzed (Participants) | 19 | 19
  Impairment of sense of taste at Day 4 | 5 | 5
  Impairment of sense of taste at Day 7: number analyzed (Participants) | 18 | 19
  Impairment of sense of taste at Day 7 | 6 | 6
  Impairment of sense of taste at Day 10: number analyzed (Participants) | 18 | 19
  Impairment of sense of taste at Day 10 | 2 | 1
  Impairment of sense of taste at Day 14: number analyzed (Participants) | 18 | 18
  Impairment of sense of taste at Day 14 | 1 | 2
  Impairment of sense of taste at Day 21: number analyzed (Participants) | 16 | 18
  Impairment of sense of taste at Day 21 | 0 | 0
  Impairment of sense of taste at Day 28: number analyzed (Participants) | 18 | 18
  Impairment of sense of taste at Day 28 | 0 | 0
  Impairment of sense of taste at Day 42: number analyzed (Participants) | 17 | 18
  Impairment of sense of taste at Day 42 | 0 | 0
  Impairment of sense of taste at Day 60: number analyzed (Participants) | 17 | 17
  Impairment of sense of taste at Day 60 | 0 | 0

3. Secondary Outcome: Sustained Improvement of Global Impression Rates
Description: Proportion of subjects in treatment group versus placebo group, respectively, who per symptom questionnaire have answered for two consecutive days: "YES" to "In the past 24 hours, have you returned to your usual health (before your COVID-19 illness)?"; "YES" to "In the past 24 hours, have you returned to your usual activities (before your COVID-19 illness)?"
Time Frame: Days 4, 7, 10, 14, 21, 28, 42, and 60 post randomization
Population: Patients reporting sustained improvement of global impression at Days 4, 7, 10, 14, 21, 28, 42, and 60
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional | Placebo
Number analyzed (Participants) | 20 | 20
Participants
  Day 4 "Returned to usual health": number analyzed (Participants) | 19 | 19
  Day 4 "Returned to usual health" | 0 | 0
  Day 7 "Returned to usual health": number analyzed (Participants) | 18 | 19
  Day 7 "Returned to usual health" | 5 | 5
  Day 10 "Returned to usual health": number analyzed (Participants) | 18 | 19
  Day 10 "Returned to usual health" | 5 | 6
  Day 14 "Returned to usual health": number analyzed (Participants) | 18 | 18
  Day 14 "Returned to usual health" | 11 | 12
  Day 21 "Returned to usual health": number analyzed (Participants) | 16 | 18
  Day 21 "Returned to usual health" | 11 | 16
  Day 28 "Returned to usual health": number analyzed (Participants) | 18 | 18
  Day 28 "Returned to usual health" | 12 | 12
  Day 42 "Returned to usual health": number analyzed (Participants) | 17 | 18
  Day 42 "Returned to usual health" | 16 | 16
  Day 60 "Returned to usual health": number analyzed (Participants) | 17 | 16
  Day 60 "Returned to usual health" | 16 | 15
  Day 4 "Returned to usual activity": number analyzed (Participants) | 19 | 19
  Day 4 "Returned to usual activity" | 0 | 4
  Day 7 "Returned to usual activity": number analyzed (Participants) | 18 | 19
  Day 7 "Returned to usual activity" | 9 | 9
  Day 10 "Returned to usual activity": number analyzed (Participants) | 18 | 19
  Day 10 "Returned to usual activity" | 11 | 15
  Day 14 "Returned to usual activity": number analyzed (Participants) | 18 | 18
  Day 14 "Returned to usual activity" | 15 | 17
  Day 21 "Returned to usual activity": number analyzed (Participants) | 16 | 18
  Day 21 "Returned to usual activity" | 15 | 17
  Day 28 "Returned to usual activity": number analyzed (Participants) | 18 | 18
  Day 28 "Returned to usual activity" | 14 | 13
  Day 42 "Returned to usual activity": number analyzed (Participants) | 17 | 18
  Day 42 "Returned to usual activity" | 16 | 17
  Day 60 "Returned to usual activity": number analyzed (Participants) | 17 | 16
  Day 60 "Returned to usual activity" | 17 | 15

4. Secondary Outcome: Time to Sustained Recovery or Resolution of Common COVID-19 Symptoms
Description: Comparison in treatment group versus placebo group, respectively, of the number of days from randomization to the first day of achieving sustained recovery and resolution rates of common COVID-19 symptoms.
Time Frame: Over 60 days post randomization
Population: The discrepancy in patient numbers (enrolled versus analyzed) is due to patients who either dropped out or have missing data.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Interventional | Placebo
Number analyzed (Participants) | 14 | 17
Days | 20.6 (18.1) | 15.4 (7.8)

5. Secondary Outcome: Time to Sustained Improvement of Global Impression
Description: Comparison in treatment group versus placebo group, respectively, of the mean number of days from randomization to the first day of achieving sustained improvement of global impression rates.
Time Frame: Over 60 days post randomization
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Interventional | Placebo
Number analyzed (Participants) | 15 | 18
Days | 10.5 (1.5) | 13.5 (2.9)

6. Secondary Outcome: Rates of Fever
Description: Proportion of subjects in treatment group versus placebo group, respectively, who, per thermometer, experienced fever at any point between enrollment and day 2 post randomization.
Time Frame: Days between enrollment and day 2 post randomization
Population: Patients who reported fever
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional | Placebo
Number analyzed (Participants) | 17 | 19
Participants | 1 | 0

7. Secondary Outcome: Oxygenation Levels
Description: Average change from baseline over 60 days in percentage of blood saturation
Time Frame: Over 60 days post randomization
Population: Patient reported oxygenation levels over 60 days.
Measure: Mean (95% Confidence Interval); unit: percentage of blood saturation
Arm/Group | Interventional | Placebo
Number analyzed (Participants) | 20 | 20
percentage of blood saturation | -0.01 [-0.01 to 0.00] | -0.01 [-0.02 to 0.01]

8. Secondary Outcome: Time in Days to Normalization of Fever and Oxygenation Levels.
Description: Comparison in treatment group versus placebo group, respectively, of the number of days from randomization to the first day of achieving sustained (i.e., at least 2 days) resolution of fever for subjects who presented with fever at any point between enrollment and day 2 post randomization; with temperature <38C or >=38C experienced in total during the first 28 days post randomization; from randomization to the first day post randomization of achieving oxygenation of SpO2>=96% in room air when resting for subjects who presented with SpO2>93% and <96% in room air, when resting, at enrollment; with oxygenation of SpO2>= 96% or SpO2>93% in room air, when resting, in total during the first 28 days post randomization.
Time Frame: 28 Days
Population: NOTE: One belnacasan participant had a fever (see outcome measure 6) which resolved on Day 4 an no placebo participants had a fever above 38C.
  NOTE: 2 placebo participants had oxygen saturation between 93 and 96% which increased to >96% on Day 7 and no belnacasan participants had an oxygen saturation below 96%.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Interventional | Placebo
Number analyzed (Participants) | 1 | 2
Days
  Time in days to normalization of fever: number analyzed (Participants) | 1 | 0
  Time in days to normalization of fever | 4 (0.00) |
  Time in days to normalization of oxygenation level: number analyzed (Participants) | 0 | 2
  Time in days to normalization of oxygenation level |  | 7 (0.00)

9. Secondary Outcome: Experiences of COVID-19 Related Deterioration and Mortality
Description: Proportion of treatment group, versus placebo group, respectively, who per subject reporting or medical records had experienced an emergency department visit, other than at study enrollment or study visits; hospitalization for COVID-19; hospitalization for COVID-19 requiring oxygen; hospitalization for COVID-19 requiring ICU; hospitalization for COVID-19 requiring ventilation; COVID-19 related death; death; hospitalization or death on Days 14, 28, and 60.
Time Frame: Days 14, 28 and 60 post randomization
Population: The number of treatment group, versus placebo group, respectively, who had COVID-related: emergency department visit, hospitalization, required oxygen, required an ICU visit, required ventilation, or died as of Days 14, 28, and 60.
Measure: Number; unit: Number of subjects
Arm/Group | Interventional | Placebo
Number analyzed (Participants) | 18 | 18
Number of subjects
  Subjects who had COVID-related: ER visit, hospitalization, ICU visit, or died by Day 14. | 0 | 0
  Subjects who had COVID-related: ER visit, hospitalization, ICU visit, or died by Day 28 | 0 | 0
  Subjects who had COVID-related: ER visit, hospitalization, ICU visit, or died by Day 60: number analyzed (Participants) | 17 | 17
  Subjects who had COVID-related: ER visit, hospitalization, ICU visit, or died by Day 60 | 0 | 0
  Subjects who required oxygen or ventilation by Day 14 | 0 | 0
  Subjects who required oxygen or ventilation by Day 28 | 0 | 0
  Subjects who required oxygen or ventilation by Day 60: number analyzed (Participants) | 17 | 17
  Subjects who required oxygen or ventilation by Day 60 | 0 | 0

10. Secondary Outcome: The Number of Subjects With COVID-19 Related Deterioration and Mortality Experiences
Description: Comparison of treatment group versus placebo group, respectively, in the number of subjects who following randomization experienced hospitalization for COVID-19 related deterioration: requiring oxygen, requiring ICU admission, requiring ventilation.
Time Frame: Over 28 days
Measure: Number; unit: participants
Arm/Group | Interventional | Placebo
Number analyzed (Participants) | 18 | 18
participants | 0 | 0

11. Secondary Outcome: Changes on the WHO 9-Point Ordinal Scale
Description: The counts of participants in the treatment group versus placebo group, respectively, who per questionnaire on WHO 9-point ordinal scale [0: Uninfected or "no clinical or virological evidence of infection"; 1: Not hospitalized, no limitations on activities; 2: Not hospitalized, limitation on activities; 3: Hospitalized, not requiring supplemental oxygen; 4: Hospitalized, requiring supplemental oxygen; 5: Hospitalized, on non-invasive ventilation or high flow oxygen devices; 6: Hospitalized, intubated; 7: Hospitalized, advanced life support including invasive mechanical ventilation or ECMO; 8: Death] had experienced an improvement from scale 2 to scale 1 or 0; an improvement from scale 1 to scale 0 ; a sustainment from scale 1 to scale 1; any improvement of the scale; any worsening of the scale; scale 4 or higher; scale 6 or higher.
Time Frame: Days 4, 7, 10, 14, 21, 28, 42, and 60 post randomization
Population: Patients reported WHO 9-point scale status from baseline to scale 1 or 0 at Days 4, 7, 10, 14, 21, 28, 42, and 60
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional | Placebo
Number analyzed (Participants) | 20 | 20
Participants
  Day 4: number analyzed (Participants) | 19 | 18
  Day 4 | 3 | 6
  Day 7: number analyzed (Participants) | 18 | 18
  Day 7 | 8 | 8
  Day 10: number analyzed (Participants) | 18 | 18
  Day 10 | 14 | 13
  Day 14: number analyzed (Participants) | 18 | 17
  Day 14 | 14 | 11
  Day 21: number analyzed (Participants) | 16 | 17
  Day 21 | 15 | 15
  Day 28: number analyzed (Participants) | 18 | 17
  Day 28 | 16 | 16
  Day 42: number analyzed (Participants) | 17 | 17
  Day 42 | 16 | 16
  Day 60: number analyzed (Participants) | 17 | 16
  Day 60 | 17 | 15

12. Secondary Outcome: Values on the WHO 9-Point Ordinal Scale
Description: Comparison of treatment group versus placebo group, respectively, in the average of daily scale value (0-8) on Days 14, 28, and 60 with respect to the number of subjects who reported as uninfected (scale value of 0), had no limitations (scale value of 1), or were experiencing limitations (scale value of 2). All patients had a score ranging between 0-2.
  A description of the WHO 9-Point Ordinal Scale follows:
  0. Uninfected or "no clinical or virological evidence of infection"
  * defined as subject answering "Yes" to "In the past 24 hours, have you returned to your usual health (before your COVID-19 illness)?"
    1. Not hospitalized, no limitations on activities
  * defined as subject answering "Yes" to "In the past 24 hours, have you returned to your usual activities (before your COVID-19 illness)?" 2. Not hospitalized, limitation on activities
  * defined as subject answering "No" to "In the past 24 hours, have you returned to your usual act
Time Frame: Days 14, 28, and 60 post randomization
Population: Subjects who reported a value from 0-2 on Days 14, 28, and 60.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interventional | Placebo
Number analyzed (Participants) | 18 | 18
units on a scale
  Average WHO-9 point scale value at Day 14 | 1.00 (0.69) | 0.94 (0.87)
  Average WHO-9 point scale value at Day 28 | 0.33 (0.69) | 0.17 (0.51)
  Average WHO-9 point scale value at Day 60: number analyzed (Participants) | 17 | 17
  Average WHO-9 point scale value at Day 60 | 0.00 (0.00) | 0.12 (0.48)

13. Secondary Outcome: Time to Improvement on the WHO 9-Point Ordinal Scale
Description: Comparison of treatment group versus placebo group, respectively, in the mean number of days from enrollment to reporting "no limitations" or "uninfected". The discrepancy in patient numbers (enrolled versus analyzed) is due to patients who either dropped out or have missing data.
Time Frame: Post treatment to Day 60
Population: Patients for whom there are data for reporting "no limitations" or "uninfected"
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Interventional | Placebo
Number analyzed (Participants) | 20 | 20
Days
  Days to "no limitations": number analyzed (Participants) | 15 | 8
  Days to "no limitations" | 9.3 (6.1) | 7.1 (5.0)
  Days to "uninfected": number analyzed (Participants) | 17 | 17
  Days to "uninfected" | 27.2 (14.3) | 19.0 (8.9)

14. Secondary Outcome: Mean Number of Days of Experiencing WHO 9-Point Ordinal Scale Values
Description: Comparison of treatment group versus placebo group, respectively, in the mean number of days on which subjects experienced "limitations", "no limitations", and "uninfected" post treatment (60 Days).
Time Frame: Post treatment through Day 60
Population: Mean number of days in which patients experienced "limitations", "no limitations" and "uninfected"
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Interventional | Placebo
Number analyzed (Participants) | 20 | 20
Days
  Limitations | 2.9 (1.8) | 2.8 (1.7)
  No limitations | 2.2 (1.9) | 1.7 (1.4)
  Uninfected | 3.0 (1.7) | 3.8 (2.1)

15. Secondary Outcome: IL-6
Description: Plasma levels of IL-6
Time Frame: Baseline and Days 7, 14, 21, 28
Population: Number of patients who had plasma IL-6 levels measured Baseline and Days 7, 14, 21, 28.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Interventional | Placebo
Number analyzed (Participants) | 20 | 20
pg/mL
  Baseline: number analyzed (Participants) | 13 | 14
  Baseline | 17.4 (13.6) | 14.6 (10.0)
  Day 7: number analyzed (Participants) | 9 | 10
  Day 7 | 15.1 (12.1) | 11.1 (8.4)
  Day 14: number analyzed (Participants) | 9 | 6
  Day 14 | 16.9 (13.4) | 9.7 (2.7)
  Day 21: number analyzed (Participants) | 5 | 7
  Day 21 | 16.0 (15.1) | 10.2 (2.1)
  Day 28: number analyzed (Participants) | 9 | 6
  Day 28 | 13.9 (10.8) | 9.7 (3.7)

16. Secondary Outcome: IL-1ra
Description: Measurement of plasma IL-1ra levels
Time Frame: Baseline and Days 7, 14, 21, 28
Population: Number of patients who had plasma IL-1ra levels measured Baseline and Days 7, 14, 21, 28.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Interventional | Placebo
Number analyzed (Participants) | 20 | 20
pg/mL
  Baseline: number analyzed (Participants) | 15 | 17
  Baseline | 37.2 (19.0) | 32.5 (14.4)
  Day 7: number analyzed (Participants) | 14 | 13
  Day 7 | 31.2 (18.1) | 26.6 (11.4)
  Day 14: number analyzed (Participants) | 12 | 11
  Day 14 | 34.0 (13.6) | 23.2 (7.7)
  Day 21: number analyzed (Participants) | 8 | 11
  Day 21 | 40.2 (14.5) | 23.7 (11.2)
  Day 28: number analyzed (Participants) | 10 | 10
  Day 28 | 37.1 (15.8) | 25.4 (7.6)

17. Secondary Outcome: IL-18
Description: Measurement of plasma levels of IL-18
Time Frame: Baseline and Days 7, 14, 21, and 28
Population: Number of patients who had plasma IL-18 levels measured Baseline and Days 7, 14, 21, 28.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Interventional | Placebo
Number analyzed (Participants) | 20 | 20
pg/mL
  Baseline: number analyzed (Participants) | 20 | 19
  Baseline | 120.1 (69.6) | 116.0 (65.9)
  Day 7: number analyzed (Participants) | 18 | 17
  Day 7 | 82.0 (60.4) | 88.6 (47.6)
  Day 14: number analyzed (Participants) | 18 | 15
  Day 14 | 77.0 (58.8) | 81.7 (38.6)
  Day 21: number analyzed (Participants) | 14 | 18
  Day 21 | 75.1 (58.9) | 80.7 (43.6)
  Day 28: number analyzed (Participants) | 16 | 17
  Day 28 | 73.7 (56.0) | 74.4 (36.6)

18. Secondary Outcome: TNF-alpha
Description: Plasma levels of TNF-alpha
Time Frame: Baseline and Days 7, 14, 21, and 28
Population: Number of patients who had plasma TNF-alpha levels measured Baseline and Days 7, 14, 21, 28.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Interventional | Placebo
Number analyzed (Participants) | 20 | 20
pg/mL
  Baseline: number analyzed (Participants) | 17 | 18
  Baseline | 131.1 (99.9) | 97.0 (46.8)
  Day 7: number analyzed (Participants) | 14 | 11
  Day 7 | 124.5 (104.2) | 97.8 (38.9)
  Day 14: number analyzed (Participants) | 13 | 12
  Day 14 | 137.1 (123.7) | 97.8 (51.4)
  Day 21: number analyzed (Participants) | 11 | 14
  Day 21 | 121.4 (112.6) | 84.0 (46.5)
  Day 28: number analyzed (Participants) | 12 | 12
  Day 28 | 128.4 (140.8) | 89.9 (42.3)

19. Secondary Outcome: Caspase-1
Description: Plasma levels of caspase-1
Time Frame: Baseline and Days 7, 14, 21, and 28
Population: Number of patients who had plasma caspase-1 levels measured Baseline and Days 7, 14, 21, 28.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Interventional | Placebo
Number analyzed (Participants) | 20 | 20
pg/mL
  Baseline: number analyzed (Participants) | 20 | 19
  Baseline | 97.2 (77.6) | 115.5 (110)
  Day 7: number analyzed (Participants) | 18 | 18
  Day 7 | 84.7 (95.2) | 104.4 (92.0)
  Day 14: number analyzed (Participants) | 18 | 17
  Day 14 | 69.5 (74.8) | 96.4 (105.8)
  Day 21: number analyzed (Participants) | 15 | 18
  Day 21 | 98.7 (120.0) | 96.4 (105.8)
  Day 28: number analyzed (Participants) | 17 | 17
  Day 28 | 101.6 (150.9) | 83.4 (66.4)

20. Secondary Outcome: Gasdermin D
Description: Plasma levels of gasdermin D
Time Frame: Baseline and Days 7, 14, 21, and 28
Population: Number of patients who had plasma gasdermin D levels measured Baseline and Days 7, 14, 21, 28.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Interventional | Placebo
Number analyzed (Participants) | 20 | 20
pg/mL
  Baseline: number analyzed (Participants) | 20 | 19
  Baseline | 2.5 (1.9) | 3.5 (2.9)
  Day 7: number analyzed (Participants) | 18 | 18
  Day 7 | 4.0 (2.5) | 4.9 (4.0)
  Day 14: number analyzed (Participants) | 18 | 17
  Day 14 | 5.0 (3.1) | 5.2 (3.6)
  Day 21: number analyzed (Participants) | 15 | 18
  Day 21 | 6.2 (3.1) | 7.2 (4.0)
  Day 28: number analyzed (Participants) | 17 | 17
  Day 28 | 5.4 (3.3) | 5.4 (2.7)

21. Secondary Outcome: G-CSF
Description: Plasma levels of G-CSF
Time Frame: Baseline and Days 7, 14, 21, and 28
Population: Number of patients who had plasma G-CSF levels measured Baseline and Days 7, 14, 21, 28.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Interventional | Placebo
Number analyzed (Participants) | 20 | 20
pg/mL
  Baseline: number analyzed (Participants) | 20 | 19
  Baseline | 137.2 (34.2) | 147.0 (56.9)
  Day 7: number analyzed (Participants) | 18 | 18
  Day 7 | 125.0 (29.1) | 106.6 (36.4)
  Day 14: number analyzed (Participants) | 18 | 17
  Day 14 | 121.4 (41.2) | 100.2 (20.8)
  Day 21: number analyzed (Participants) | 15 | 18
  Day 21 | 114.5 (34.9) | 103.8 (21.3)
  Day 28: number analyzed (Participants) | 16 | 17
  Day 28 | 122.5 (45.3) | 102.9 (24.1)

ADVERSE EVENTS:
Time Frame: From the time of enrollment through Day 60
Arm/Group | Interventional | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 0/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventional (N=20) | Placebo (N=20)
Chest pain (Cardiac disorders) | 2 (2) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT05164120/Prot_SAP_000.pdf